CLINICAL TRIAL: NCT00158197
Title: Behavior Change: Reinforcement Schedule Effects
Brief Title: Long-term Behavior Change - 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friends Research Institute, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-17407-1; R01DA017407 (NIH); R01-17407-1
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Amphetamine-related Disorders
Keywords: Adherence; Amphetamine-Related Disorders; Behavior Therapy; Contingency management; Drug Counseling; health behaviors; methamphetamine; sexual risk behaviors; substance dependence
MeSH Terms: conditions — Amphetamine-Related Disorders; Health Behavior; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- continuous voucher schedule (Experimental): Those in the continuous condition will receive a contingency management voucher each time they test negative for methamphetamine. The initial voucher value will be $2.50. Each consecutive instance of abstinence will increase the magnitude of the voucher by $1.50. Three consecutive abstinences will result in the delivery of a $10.00 bonus. Provision of a methamphetamine-positive urine sample, or failure to test, will result in a reset in the voucher magnitude back to its original level from whence the progression can begin again. All participants will provide observed urine samples three times a week (e.g., M, W, & F) for twelve weeks and will complete study-related measures one time per week.
  Interventions: Behavioral: contingency management voucher
- intermittent predictable schedule (Experimental): Those in the intermittent predictable condition will earn a contingency management voucher when they provide three consecutive methamphetamine-negative urine tests. Participants in the intermittent predictable condition will receive $22.00 for the provision of their first three consecutive methamphetamine-negative urine samples, $35.50 for the provision of their second set of three consecutive instances of methamphetamine-negative urine samples, and so forth. There are no bonuses for consecutive instances of abstinence in the intermittent predictable condition. Provision of a methamphetamine-positive urine sample, or failure to test, will result in a reset in the voucher magnitude back to its original level from whence the progression can begin again. All participants will provide observed urine samples three times a week (e.g., M, W, & F) for twelve weeks and will complete study-related measures one time per week.
  Interventions: Behavioral: contingency management voucher
- intermittent unpredictable schedule (Experimental): Those in the intermittent unpredictable condition will be eligible to receive a contingency management voucher on one day a week. Participants in this group will receive a voucher for $22.00 following their first 3 methamphetamine-negative urine tests. They will then be eligible to receive a voucher one day a week if all of their urine tests since the receipt of their last voucher were methamphetamine negative. They will receive a voucher for $35.50 for the provision of their second set of 3 consecutive instances of methamphetamine-negative urine samples, $49.00 for their third set of 3 consecutive instances, and so forth. The day of the week on which the voucher will be available will be randomly selected for each week and the participants will not know which day of the week they will be eligible to receive a voucher until they have provided their urine test. All participants will provide observed urine samples M, W, & F for 12 wks and complete measures 1x/wk.
  Interventions: Behavioral: contingency management voucher
- standard (No Intervention): Participants assigned to the standard condition will not receive vouchers for the provision of clean urines. All participants will provide observed urine samples three times a week (e.g., M, W, & F) for twelve weeks and will complete study-related measures one time per week.

INTERVENTIONS:
Behavioral: contingency management voucher — participants receive vouchers for the provision of methamphetamine-negative urines. Vouchers can be redeemed for goods and services compatible with non-drug using behaviors.
  Arms: continuous voucher schedule; intermittent predictable schedule; intermittent unpredictable schedule

SUMMARY:
The purpose of this study is to determine if different reinforcement procedures (i.e., schedules) produce different patterns of long-term abstinence from methamphetamine. We anticipate that the three contingency management conditions will promote longer periods of abstinence in the year following treatment relative to the standard control group. Furthermore, we predict that the intermittent reinforcement procedures will produce longer periods of continued abstinence (i.e., long-term behavior change) in the year following treatment than the continuous reinforcement procedure. Finally, we predict that the intermittent unpredictable schedule will produce longer lasting behavior change than the intermittent predictable schedule. Methamphetamine use will be measured using urine toxicology and self-report of methamphetamine use.

DETAILED DESCRIPTION:
Briefly the four study conditions are: (1) standard treatment which consists of 16 weeks of psychosocial treatment, (2) continuous contingency management which consists of 16 weeks of psychosocial treatment with a contingency management procedure in effect during the first twelve weeks in which vouchers are made available after each provision of a methamphetamine-negative urine test, (3) intermittent predictable contingency management which consists of 16 weeks of psychosocial treatment with a contingency management procedure in effect during the first twelve weeks in which vouchers are available after the provision of every three consecutive methamphetamine-negative urine samples, and (4) intermittent unpredictable contingency management which consists of 16 weeks of psychosocial treatment with a contingency management procedure in effect during the first twelve weeks in which vouchers are available on one day each week (randomly selected after the first week) for the provision of methamphetamine-negative urine samples provided all urine samples since delivery of the last reinforcer were also methamphetamine negative.

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for methamphetamine dependence
* Willing and able to comply with study procedures
* Willing and able to provide written informed consent

Exclusion Criteria:

* Have a medical condition that, in the study Principal Investigator (PI's) judgment, might interfere with safe study participation
* Have a recent (past 30 days) history of suicide attempts and/or current serious suicidal intention or plan as assessed by the Beck Depression Inventory (BDI)
* Have a history of violent criminal behavior or be on parole
* Any other circumstances that, in the opinion of the PI, would interfere with safe study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2004-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Roll, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Friends Research Institute, Los Angeles, California
  - Friends Research Institute, Rancho Cucamonga, California

REFERENCES:
- [Result] Roll JM, Chudzynski J, Cameron JM, Howell DN, McPherson S. Duration effects in contingency management treatment of methamphetamine disorders. Addict Behav. 2013 Sep;38(9):2455-62. doi: 10.1016/j.addbeh.2013.03.018. Epub 2013 Apr 3. PMID 23708468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and enrollment began in January 2005 and ended . Individuals were recruited from the community via radio and newspaper ads, flyers, and word of mouth.
Pre-assignment Details: The main reasons individuals were excluded from the trial prior to group assignment was not meeting inclusion criteria and discontinuing treatment prior to randomization.
Groups:
- Intermittent Predictable Schedule: Those in the intermittent predictable condition earned a voucher when they provide three consecutive methamphetamine-negative urine tests. Participants in the intermittent predictable condition received $22.00 for the provision of their first three consecutive methamphetamine-negative urine samples, $35.50 for the provision of their second set of three consecutive instances of methamphetamine-negative urine samples, and so forth. There were no bonuses for consecutive instances of abstinence in the intermittent predictable condition. Provision of a methamphetamine-positive urine sample, or failure to test, resulted in a reset in the voucher magnitude back to its original level from whence the progression can begin again.
  contingency management voucher : participants receive vouchers for the provision of methamphetamine-negative urines. Vouchers can be redeemed for goods and services compatible with non-drug using behaviors.
- Continuous Schedule: Those in the continuous condition received a voucher each time they tested negative for methamphetamine. The initial voucher value was $2.50. Each consecutive instance of abstinence increased the magnitude of the voucher by $1.50. Three consecutive abstinences resulted in the delivery of a $10.00 bonus. Provision of a methamphetamine-positive urine sample, or failure to test, resulted in a reset in the voucher magnitude back to its original level from whence the progression could begin again.
  contingency management voucher : participants receive vouchers for the provision of methamphetamine-negative urines. Vouchers can be redeemed for goods and services compatible with non-drug using behaviors.
- Intermittent Unpredictable Schedule: Participants in the unpredictable intermittent condition earned vouchers of the same magnitude as those in the predictable intermittent condition and at approximately the same rate (i.e., $22.00 for the provision of their first three consecutive methamphetamine-negative urine samples, $35.50 for the provision of their second week of methamphetamine-negative urines, etc). More specifically, participants in this group received a voucher for $22.00 following their first three methamphetamine-negative urine tests. Following that they were eligible to receive a voucher one day a week if all of their urine tests since the receipt of their last voucher were methamphetamine negative. This date was randomly determined and they did not know in advance what day it was.
  contingency management voucher : participants receive vouchers for the provision of methamphetamine-negative urines. Vouchers can be redeemed for goods and services compatible with non-drug using behaviors.
- Standard: Participants assigned to the standard condition did not receive vouchers for the provision of clean urines.
Period: Overall Study
Arm/Group | Intermittent Predictable Schedule | Continuous Schedule | Intermittent Unpredictable Schedule | Standard
Started | 32 | 30 | 28 | 29
Completed | 32 | 30 | 28 | 29
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intermittent Predictable Schedule: Those in the intermittent predictable condition will earn a voucher when they provide three consecutive methamphetamine-negative urine tests. Participants in the intermittent predictable condition will receive $22.00 for the provision of their first three consecutive methamphetamine-negative urine samples, $35.50 for the provision of their second set of three consecutive instances of methamphetamine-negative urine samples, and so forth. There are no bonuses for consecutive instances of abstinence in the intermittent predictable condition. Provision of a methamphetamine-positive urine sample, or failure to test, will result in a reset in the voucher magnitude back to its original level from whence the progression can begin again.
  contingency managment voucher : participants receive vouchers for the provision of methamphetamine-negative urines. Vouchers can be redeemed for goods and services compatible with non-drug using behaviors.
- Continuous Voucher Schedule: Those in the continuous condition will receive a voucher each time they test negative for methamphetamine. The initial voucher value will be $2.50. Each consecutive instance of abstinence will increase the magnitude of the voucher by $1.50. Three consecutive abstinences will result in the delivery of a $10.00 bonus. Provision of a methamphetamine-positive urine sample, or failure to test, will result in a reset in the voucher magnitude back to its original level from whence the progression can begin again.
  contingency managment voucher : participants receive vouchers for the provision of methamphetamine-negative urines. Vouchers can be redeemed for goods and services compatible with non-drug using behaviors.
- Intermittent Unpredictable Schedule: Those in the intermittent unpredictable condition will be eligible to receive a voucher on one day a week. This date will be randomly determined and they will not know in advance what day it will be. Participants in this group will receive a voucher following their first three methamphetamine-negative urine tests. Following that they will be eligible to receive a voucher one day a week if all of their urine tests since the receipt of their last voucher were methamphetamine negative. The day of the week on which the voucher will be available will be randomly selected for each week and the participants will not know which day of the week they will be eligible to receive a voucher until they have provided their urine test.
  contingency managment voucher : participants receive vouchers for the provision of methamphetamine-negative urines. Vouchers can be redeemed for goods and services compatible with non-drug using behaviors.
- Standard: Participants assigned to the standard condition will not receive vouchers for the provision of clean urines.
- Total: Total of all reporting groups
Arm/Group | Intermittent Predictable Schedule | Continuous Voucher Schedule | Intermittent Unpredictable Schedule | Standard | Total
Number analyzed (Participants) | 32 | 30 | 28 | 29 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 32 | 30 | 28 | 29 | 119
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (8.2) | 32.5 (10) | 30.3 (10.9) | 24.8 (10.1) | 32 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 13 | 14 | 50
  Male | 19 | 20 | 15 | 15 | 69
Region of Enrollment [Number; unit: participants]
  United States | 32 | 30 | 28 | 29 | 119

OUTCOME MEASURES:

1. Primary Outcome: Methamphetamine Use During Intervention
Description: Drug use measured by urine toxicology conducted by on site Enzyme-multiplied immunoassay technique (EMIT) assay over time.
Time Frame: 3x/week for 16 weeks
Population: All individuals randomized were included in the analysis (i.e., intention to treat).
Measure: Number; unit: percentage of negative urine samples
Units Other Than Participants: Urine samples
Groups:
- Intermittent Predictable Schedule: Those in the intermittent predictable condition will earn a voucher when they provide three consecutive methamphetamine-negative urine tests. Participants in the intermittent predictable condition will receive $22.00 for the provision of their first three consecutive methamphetamine-negative urine samples, $35.50 for the provision of their second set of three consecutive instances of methamphetamine-negative urine samples, and so forth. There are no bonuses for consecutive instances of abstinence in the intermittent predictable condition. Provision of a methamphetamine-positive urine sample, or failure to test, will result in a reset in the voucher magnitude back to its original level from whence the progression can begin again.
  contingency management voucher : participants receive vouchers for the provision of methamphetamine-negative urines. Vouchers can be redeemed for goods and services compatible with non-drug using behaviors.
- Continuous Voucher Schedule: Those in the continuous condition will receive a voucher each time they test negative for methamphetamine. The initial voucher value will be $2.50. Each consecutive instance of abstinence will increase the magnitude of the voucher by $1.50. Three consecutive abstinences will result in the delivery of a $10.00 bonus. Provision of a methamphetamine-positive urine sample, or failure to test, will result in a reset in the voucher magnitude back to its original level from whence the progression can begin again.
  contingency management voucher : participants receive vouchers for the provision of methamphetamine-negative urines. Vouchers can be redeemed for goods and services compatible with non-drug using behaviors.
- Intermittent Unpredictable Schedule: Those in the intermittent unpredictable condition will be eligible to receive a voucher on one day a week. This date will be randomly determined and they will not know in advance what day it will be. Participants in this group will receive a voucher following their first three methamphetamine-negative urine tests. Following that they will be eligible to receive a voucher one day a week if all of their urine tests since the receipt of their last voucher were methamphetamine negative. The day of the week on which the voucher will be available will be randomly selected for each week and the participants will not know which day of the week they will be eligible to receive a voucher until they have provided their urine test.
  contingency management voucher : participants receive vouchers for the provision of methamphetamine-negative urines. Vouchers can be redeemed for goods and services compatible with non-drug using behaviors.
Arm/Group | Intermittent Predictable Schedule | Continuous Voucher Schedule | Intermittent Unpredictable Schedule | Standard
Number analyzed (Participants) | 32 | 30 | 28 | 29
Number analyzed (Urine samples) | 1536 | 1440 | 1344 | 1392
percentage of negative urine samples | 65.17 | 60.35 | 57.74 | 42.81
Statistical Analysis 1: Comparison: Continuous Voucher Schedule vs Standard; Test type: Superiority or Other; p < 0.01, Generalized estimating equations; Odds Ratio (OR) = 1.98 — Value represents the odds of submitting a methamphetamine negative urine sample in the treatment group (1 of 3) compared to the standard care group
Statistical Analysis 2: Comparison: Intermittent Predictable Schedule vs Standard; Test type: Superiority or Other; p < 0.01, Generalized estimating equations; Odds Ratio (OR) = 2.40 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Intermittent Unpredictable Schedule vs Standard; Test type: Superiority or Other; p < 0.01, Generalized estimating equations; Odds Ratio (OR) = 1.72 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Methamphetamine Use, Measured by Number of Consecutive Days of Abstinence
Description: Drug use measured by urine toxicology conducted by on site EMIT assay and added up to obtain how many days of consecutive abstinence were observed for each individual
Time Frame: 16 Weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intermittent Predictable Schedule | Continuous Voucher Schedule | Intermittent Unpredictable Schedule | Standard
Number analyzed (Participants) | 32 | 30 | 28 | 29
days | 22.42 (15.36) | 22.7 (17.60) | 20.32 (18.64) | 11.10 (12.58)
Statistical Analysis 1: Comparison: Intermittent Predictable Schedule vs Continuous Voucher Schedule vs Intermittent Unpredictable Schedule vs Standard; Test type: Superiority or Other; p = 0.02, ANOVA — Yes, the a priori plan to handle post hoc multiple comparisons was to use the method of Bonferroni adjustment. Thus, the new alpha level for these comparisons was <0.0125
Statistical Analysis 2: Comparison: Intermittent Predictable Schedule vs Standard; Test type: Superiority or Other; p < 0.01, t-test, 2 sided
Statistical Analysis 3: Comparison: Continuous Voucher Schedule vs Standard; Test type: Superiority or Other; p < 0.01, t-test, 2 sided
Statistical Analysis 4: Comparison: Intermittent Unpredictable Schedule vs Standard; Test type: Superiority or Other; p = 0.20, t-test, 2 sided

3. Primary Outcome: Methamphetamine Use, Follow-Up
Description: Drug use measured by urine toxicology conducted by on site EMIT assay over time
Time Frame: 1x/month for 4 months
Measure: Number; unit: percentage of negative urine samples
Units Other Than Participants: Urine samples
Arm/Group | Intermittent Predictable Schedule | Continuous Voucher Schedule | Intermittent Unpredictable Schedule | Standard
Number analyzed (Participants) | 32 | 30 | 28 | 29
Number analyzed (Urine samples) | 128 | 120 | 112 | 116
percentage of negative urine samples | 90.79 | 88.89 | 88.62 | 87.30
Statistical Analysis 1: Comparison: Intermittent Unpredictable Schedule vs Standard; We used GEE to investigate change in methamphetamine abstinence (i.e., provision of a negative methamphetamine UA) during the follow-up period; Test type: Superiority or Other; p = 0.78, Generalized estimating equations
Statistical Analysis 2: Comparison: Continuous Voucher Schedule vs Standard; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.68, Generalized estimating equations
Statistical Analysis 3: Comparison: Intermittent Predictable Schedule vs Standard; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.20, Generalized estimating equations

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected at each study and follow-up visit, for 1 year.
Arm/Group | Continuous Voucher Schedule | Intermittent Predictable Schedule | Intermittent Unpredictable Schedule | Standard
Serious Adverse Events (participants affected / at risk) | 5/119 | 3/119 | 1/119 | 1/119
Other Adverse Events (participants affected / at risk) | 1/119 | 5/119 | 1/119 | 3/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Voucher Schedule (N=119) | Intermittent Predictable Schedule (N=119) | Intermittent Unpredictable Schedule (N=119) | Standard (N=119)
slipped vertebral disk (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Pain and stiffness in neck.Diagnosed with a slipped vertebral disk and underwent surgery to correct it. Ct was prescribed painkillers and assigned physical therapy.
back and lung injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Ct hospitalized for stab wounds in the face and back. Ct underwent surgery for back and lung injuries. Ct was released with prescriptions for painkillers, iron and glucose.
child birth (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Ct reported seeking medical attention due to labor pains. Ct gave birth to health child.
pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Ct hospitalized for difficulty breathing and edema, diagnosed with pneumonia. Ct was hospitalized and received fluids and antibiotics intravenously along with oxygen and breathing treatments.
chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Ct hospitalized to monitor chest pain and tightness. Prescribed heart and pain medication.
Diabetes Mellitus, Type II (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Client sought medical attention due to increased thirst and frequency in urination. Client was hospitalized overnight to monitor glucose levels. Client was diagnosed with Diabetes Mellitus, Type II.
High glucose levels (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Client sought medical attention for frequent urination and thirst. Client admitted to hospital for high glucose levels and was given insulin for stabilization.
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Client sought medical attention due to pains in chest and difficulty breathing. Client was diagnosed with pneumonia.
breathing difficulty (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Client sought medical attention as he was having difficulty breathing hearing properly. Client diagnosed with infection that progressed due to high blood sugar levels.
nerve pain (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Client underwent surgery to alleviate compression of the seventh cranial nerve.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Voucher Schedule (N=119) | Intermittent Predictable Schedule (N=119) | Intermittent Unpredictable Schedule (N=119) | Standard (N=119)
eye surgery (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Ct reported undergoing surgery on left eye to remove cataract. Ct was released the same day with a prescription for steroid eye drops.
lower back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Ct sought medical attention for lower back pain. Ct was diagnosed with pinched sciatic nerve, herniated disc, low back muscle strain, and lumbar muscle strain.
abscesses on legs (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Ct reported seeking medical attention for abscesses on legs. Ct underwent minor surgery to remove boils, and was released the same day.
rash and blisters (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Ct sought medical attention for rashes and blisters on both legs, which spread throughout body. Ct prescribed broad-spectrum antibiotics, antivirals, and topical ointments
fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Ct reported receiving medical attention for a high fever. Ct was diagnosed with a kidney infection, prescribed an antibiotic, and released the same day.
decayed teeth (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) — Client reported receiving oral surgery for decayed teeth. Ct was released the same day with antibiotics.
pain and swelling (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Client sought medical attention for pain and swelling in testicular area. Ct was diagnosed with build-up of fluid. Client to schedule procedure for drainage.
eye lesions (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Client sought medical attention for eye lesions. Ct was diagnosed with Herpes of the eyes, and was prescribed antibiotic ointments and antiviral drops.
tooth pain (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Ct reported seeking medical attention for tooth pain. Ct told to schedule tooth extractions.
leg injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Ct sought medical attention due to a leg injury as a result of falling while hiking. Ct received 21 stitches in left leg, and was prescribed antibiotics.
broken thumb (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Client reported seeking medical attention for broken thumb. Splint was placed on client's thumb

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No